CLINICAL TRIAL: NCT07177300
Title: Effectiveness of Nontraditional Hydroxyurea Algorithms: Novel and Clinical Evaluations (ENHANCE)
Acronym: ENHANCE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Greater Cincinnati Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENHANCE; GCF_Quinn (Other Grant/Funding Number: Greater Cinti Foundation)
Record Dates: First submitted 2025-08-18; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Anemia (HbSS); Sickle-β0-thalassemia (HbSβ0)
Keywords: sickle cell anemia; SCD; sickle cell; hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Aging; Pharmacogenomic Variants; Maximum Tolerated Dose

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single-arm therapeutic trial of pharmacokinetics (PK)-optimized oral hydroxyurea at maximum tolerated dose (MTD) for the treatment of sickle cell anemia (SCA) with long-term follow-up.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Observational Treatment Group (Single Arm) (Experimental): All children with sickle cell anemia who are started on hydroxyurea for clinical indicators between 6 months and 5 years of age can do so on this observational study with PK-optimized hydroxyurea dosing.
  Interventions: Drug: PK-optimized oral hydroxyurea at MTD until 15 years of age.

INTERVENTIONS:
Drug: PK-optimized oral hydroxyurea at MTD until 15 years of age. — Because people are different, we will measure how each participant's body absorbs and eliminates the medicine, hydroxyurea, using blood tests. This information will be used to determine the best dose for each participant (rather than using the same weight-based dose for everyone).
  Other Names: pharmacokinetic; maximum tolerated dose

SUMMARY:
The main reason for this research study is to learn more about hydroxyurea and the treatment of sickle cell anemia (SCA). Hydroxyurea is a medication that has been studied for many years and has been shown to provide benefits for people with SCA.

In this research study, the investigators hope to learn more about how to improve the dosing and monitoring of hydroxyurea and learn more about the long-term effects of hydroxyurea over time. Hydroxyurea is usually dosed based only on your weight. Our study will use a new way to select a starting dose that is based on how each patient absorbs hydroxyurea.

DETAILED DESCRIPTION:
The EHANCE study will address key knowledge gaps about hydroxyurea for young children with SCA in nine innovative ways:

* Novel functional assessments of brain, heart, kidneys, spleen, and eyes to assess organ protection in young children who receive hydroxyurea at MTD;
* State-of-the-art assays to assess the benefits of hydroxyurea on growth, development, and reproductive health into puberty including serial measurements of pubertal development and sex hormones;
* A simplified PK-guided strategy to optimize hydroxyurea initiation and dosing, with a long-term goal of validating pharmacogenomic approaches to expand treatment and achieve sustained HbF induction;
* A novel single-cell quantitative HbF/F-cell assay, developed utilizing imaging flow cytometry, will determine the distribution of HbF/F-cell across all F-cells, rather than simply estimating the mean value of HbF/F-cell;
* Collection of genomic DNA samples to allow serial quantitation of clonal hematopoiesis in treated children, to evaluate the possibility for potential emergence of clones with an increased risk of leukemic transformation;
* Studies on primary erythroblasts freshly isolated from patients and control subjects with single cell multiome analysis to evaluate in vivo cis and trans-acting elements that regulate HbF and how they are affected by hydroxyurea;
* Evaluation of cellular mechanisms by which hydroxyurea at MTD can regularly achieve >30% HbF with near-pancellular distribution, similar to levels currently touted with 'curative' gene therapy regimens;
* Exploration of the benefits of early hydroxyurea treatment initiation, in terms of γ-globin de-repression to optimize HbF induction, through unknown cellular mechanisms that may be developmentally regulated.

  3. SPECIFIC AIMS Aim 1: Document the long-term benefits and risks of long-term hydroxyurea treatment at MTD.

Aim 2: Perform pharmacokinetic (PK) and pharmacodynamic (PD) assessment of hydroxyurea at MTD.

Aim 3: Investigate the cellular mechanisms by which hydroxyurea leads to induction of protective HbF and how timing of treatment initiation and dose optimization affect the efficacy of this process.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell anemia (HbSS) or sickle-β0-thalassemia (HbSβ0)
* Age 6 months at the time of enrollment
* Clinical decision by patient, family, and healthcare provider to initiate hydroxyurea therapy

Exclusion Criteria:

* Current treatment with regularly scheduled blood transfusions
* Sickle-hemoglobin C disease (HbSC), sickle-β+-thalassemia (HbSβ+)

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Composite Organ Injury | Through study completion, an average of 10 years
  Evidence of injury in any of four critical organ systems: brain, kidney, heart, or spleen. Participants will be classified as having met the composite endpoint if they fulfill at least one of the organ-specific criteria listed: cerebral infarction (silent or overt) or steno-occlusive vasculopathy by MRI of brain; urine albumin-to-creatinine ratio (UACR) > 300 mg/g; extracellular volume fraction (ECV) > 0.35 on cardiac MRI; or erythrocyte pit count < 5%

SECONDARY OUTCOMES:
longitudinal change in fetal hemoglobin percentage (HbF%) | Through study completion, an average of 10 years
  HbF is a well-established mechanistic surrogate marker in SCA that is strongly associated with reduced sickling and organ injury across multiple organ systems. This endpoint will quantify the sustained biological effectiveness of early PK-guided hydroxyurea dosing.
Longitudinal change in hemoglobin concentration (g/dL) | Through study completion, an average of 10 years.
  A beneficial laboratory response to hydroxyurea would include less severe anemia (measured by hemoglobin concentration). This is reported in a complete blood count (CBC).
Longitudinal change in reticulocyte count (10^9/L) | Through study completion, an average of 10 years.
  A beneficial laboratory response to hydroxyurea would include a decreased reticulocyte count, indicating less severe anemia. This is reported with a complete blood count (CBC).
Longitudinal change in absolute neutrophil count (10^9/L) | Through study completion, an average of 10 years.
  A surrogate marker of hydroxyurea effectiveness and adherence is the absolute neutrophil count (ANC). Hydroxyurea is titrated according to the ANC. This is reported in a complete blood count (CBC) with differential leukocyte count.
Longitudinal change in mean cell volume (fL) | Through study completion, an average of 10 years.
  A surrogate marker of hydroxyurea effectiveness and adherence is the mean cell volume (MCV). This is reported in a complete blood count (CBC).
F-cell fraction (%) | Through study completion, an average of 10 years.
  Flow cytometric determination of the fraction of HbF-containing red blood cells (F-cells).
Adverse events | Through study completion, an average of 10 years.
  The occurrence of adverse events while on study will be continually monitored and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Charles T. Quinn, Professor of Pediatrics, M.D., M.S., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hay SB, Ferchen K, Chetal K, Grimes HL, Salomonis N. The Human Cell Atlas bone marrow single-cell interactive web portal. Exp Hematol. 2018 Dec;68:51-61. doi: 10.1016/j.exphem.2018.09.004. Epub 2018 Sep 21. PMID 30243574
- [Background] Marahatta A, Megaraj V, McGann PT, Ware RE, Setchell KD. Stable-Isotope Dilution HPLC-Electrospray Ionization Tandem Mass Spectrometry Method for Quantifying Hydroxyurea in Dried Blood Samples. Clin Chem. 2016 Dec;62(12):1593-1601. doi: 10.1373/clinchem.2016.263715. Epub 2016 Sep 30. PMID 27694393
- [Background] Vassiliou G. Telomere Length and Clonal Hematopoiesis. N Engl J Med. 2023 Jun 29;388(26):2481-2484. doi: 10.1056/NEJMe2303022. Epub 2023 May 4. No abstract available. PMID 37140164
- [Background] Bowman RL, Busque L, Levine RL. Clonal Hematopoiesis and Evolution to Hematopoietic Malignancies. Cell Stem Cell. 2018 Feb 1;22(2):157-170. doi: 10.1016/j.stem.2018.01.011. PMID 29395053
- [Background] Sankaran VG, Xu J, Orkin SH. Advances in the understanding of haemoglobin switching. Br J Haematol. 2010 Apr;149(2):181-94. doi: 10.1111/j.1365-2141.2010.08105.x. Epub 2010 Mar 1. PMID 20201948
- [Background] Ware RE, Davis BR, Schultz WH, Brown RC, Aygun B, Sarnaik S, Odame I, Fuh B, George A, Owen W, Luchtman-Jones L, Rogers ZR, Hilliard L, Gauger C, Piccone C, Lee MT, Kwiatkowski JL, Jackson S, Miller ST, Roberts C, Heeney MM, Kalfa TA, Nelson S, Imran H, Nottage K, Alvarez O, Rhodes M, Thompson AA, Rothman JA, Helton KJ, Roberts D, Coleman J, Bonner MJ, Kutlar A, Patel N, Wood J, Piller L, Wei P, Luden J, Mortier NA, Stuber SE, Luban NLC, Cohen AR, Pressel S, Adams RJ. Hydroxycarbamide versus chronic transfusion for maintenance of transcranial doppler flow velocities in children with sickle cell anaemia-TCD With Transfusions Changing to Hydroxyurea (TWiTCH): a multicentre, open-label, phase 3, non-inferiority trial. Lancet. 2016 Feb 13;387(10019):661-670. doi: 10.1016/S0140-6736(15)01041-7. Epub 2015 Dec 6. PMID 26670617
- [Background] Hankins JS, Helton KJ, McCarville MB, Li CS, Wang WC, Ware RE. Preservation of spleen and brain function in children with sickle cell anemia treated with hydroxyurea. Pediatr Blood Cancer. 2008 Feb;50(2):293-7. doi: 10.1002/pbc.21271. PMID 17554794
- [Background] Letvin NL, Linch DC, Beardsley GP, McIntyre KW, Nathan DG. Augmentation of fetal-hemoglobin production in anemic monkeys by hydroxyurea. N Engl J Med. 1984 Apr 5;310(14):869-73. doi: 10.1056/NEJM198404053101401. PMID 6199670
- [Background] Platt OS. Hydroxyurea for the treatment of sickle cell anemia. N Engl J Med. 2008 Mar 27;358(13):1362-9. doi: 10.1056/NEJMct0708272. No abstract available. PMID 18367739
- [Background] Ware RE. Optimizing hydroxyurea therapy for sickle cell anemia. Hematology Am Soc Hematol Educ Program. 2015;2015:436-43. doi: 10.1182/asheducation-2015.1.436. PMID 26637755
- [Background] Lanzkron S, Carroll CP, Haywood C Jr. Mortality rates and age at death from sickle cell disease: U.S., 1979-2005. Public Health Rep. 2013 Mar-Apr;128(2):110-6. doi: 10.1177/003335491312800206. PMID 23450875
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Vichinsky E, Hurst D, Earles A, Kleman K, Lubin B. Newborn screening for sickle cell disease: effect on mortality. Pediatrics. 1988 Jun;81(6):749-55. PMID 3368274